CLINICAL TRIAL: NCT05063903
Title: Assessment of Exercise Capacity in Single-ventricle Patients Undergoing Fontan Procedure
Brief Title: Exercise Capacity in Patients With Fontan Procedure
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Haluk TEKERLEK, Principal Investigator/Research Assistant, Hacettepe University
Other Study IDs: exercisecapacityfontan
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Single-ventricle; Fontan Procedure
Keywords: Exercise capacity; Six minute walk test; Incremental shuttle walk test; Fontan procedure
MeSH Terms: conditions — Univentricular Heart | interventions — Demography; Hand Strength; Body Composition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan Group: Fontan Group Inclusion Criteria
  be between the ages of 8-50 Having undergone Fontan operation in our hospital or another center Clinical stability of the patients (preserved ventricular function), No change in ongoing drug therapy that adversely affects clinical stability, At least 1 year after the operation and to be followed in the Pediatric Cardiology Polyclinic of our hospital
  Fontan Group Exclusion Criteria:
  Inability to access the patient's medical data Neurological and/or genetic musculoskeletal disease Having orthopedic and cognitive problems that prevent testing The patient's and/or family's unwillingness to participate in the study
  Interventions: Other: Demographic and clinical characteristics, incremental shuttle walk test, six minute walk test, hand grip strength, M. Quadriceps isometric muscle strength, body composition
- Control Group: Control Group Inclusion Criteria:
  Not have cardiovascular, neurological and/or genetic musculoskeletal disease Not having orthopedic and cognitive problems that prevent testing The patient's and/or family's willingness to participate in the study
  Interventions: Other: Demographic and clinical characteristics, incremental shuttle walk test, six minute walk test, hand grip strength, M. Quadriceps isometric muscle strength, body composition

INTERVENTIONS:
Other: Demographic and clinical characteristics, incremental shuttle walk test, six minute walk test, hand grip strength, M. Quadriceps isometric muscle strength, body composition — Demographic and clinical characteristics Age and complaints, post-operative follow-up, other problems, medications, ECHO and ECG findings, laboratory tests (complete blood count, liver and kidney function tests, brain natriuretic peptide (BNP) level)
  Hand grip strength Right and left hand grip strength the highest of the three measurements
  Lower extremity muscle strength Maximum isometric muscle strength of the quadriceps femoris
  Body composition Body fat ratio, lean body weight and fat weight by bioelectrical impedance analysis
  6 minute walk test The six minute walk test distance recorded in meters
  Incremental shuttle walk test The lap number, the number of laps of the last level they can reach, and the walking/running distances recorded in meters

SUMMARY:
In literature, it has been reported that exercise capacity decreases in single-ventricle patients undergoing Fontan Procedure due to various factors related to surgery and underlying cardiac anomaly. Cardiopulmonary exercise test (CPET) was generally used to evaluate exercise capacity in children and adults with fontan circulation. The fact that CPET requires a clinically expert team and equipment and is more expensive does not always make it possible to perform routine cardiopulmonary exercise testing. In some cases, field tests evaluating submaximal and maximal exercise capacity may be more practical than cardiopulmonary exercise testing. Therefore, in this study, it is aimed to evaluate the exercise capacity of Fontan patients with 6-minute walking test and incremental shuttle walk test and to compare vital signs during the tests.

ELIGIBILITY:
Fontan Group Inclusion Criteria

* be between the ages of 8-50
* Having undergone Fontan operation in our hospital or another center
* Clinical stability of the patients (preserved ventricular function),
* No change in ongoing drug therapy that adversely affects clinical stability,
* At least 1 year after the operation and to be followed in the Pediatric Cardiology Polyclinic of our hospital

Fontan Group Exclusion Criteria:

* Inability to access the patient's medical data
* Neurological and/or genetic musculoskeletal disease
* Having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's unwillingness to participate in the study

Control Group Inclusion Criteria:

* Not have cardiovascular, neurological and/or genetic musculoskeletal disease
* Not having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's willingness to participate in the study

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The number of individuals to be included in the study was determined as 27 According to the power analysis at α=0.05 and β=0.20 (for 80% power). In this study, the medical information and medical records of the patients (patient files, computer records, etc.) will be examined and recorded. Patients aged 8-50 years who underwent the fonton procedure and were followed by Hacettepe University, Department of Pediatric Cardiology will be included in the study. The eligible patients will be referred to Faculty of Physical Therapy and Rehabilitation after the routine evaluations are completed. Control cases planned to be included in the study to be compared with the results of Fontan patients will be created by inviting the healthy relatives of the patients who applied to our faculty to participate in the study. In addition, control cases will be invited to work through an online advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Incremental shuttle walk test distance | 30-45 minutes
  For the incremental shuttle walk test, it will be adjusted to a total of 10 meters with 2 cones placed at a distance of 9.0 meters from each other and a rotational margin of 0.5 meters. In this system, the patient will be asked to walk in a round-trip way by adapting to the increasing speed and the sound coming from outside. Walking/running distances of the patients in meters will be recorded.
6 minute walk test distance | 15-20 minutes
  The standard test protocol will be applied in a continuous 30 meter corridor. The patient wearing comfortable clothes and shoes will be given standard instructions and verbal guidance during the test. The distance the patient walked during the test will be recorded in meters.
Right and left hand grip strength | 15-20 minutes
  Right and left hand grip strength will be measured using a hand grip strength hand dynamometer (Jamar, Sammons Preston, Rolyon, Bolingbrook, IL, USA). Measurements shall be made using standard procedures, right and left sides, with the arms at the side of the trunk, the elbow in a 90 degree flexion position, and the forearm and wrist in a neutral position. The highest of the three measurements will be considered as hand grip strength
Maximum isometric muscle strength of the quadriceps femoris | 15-20 minutes
  The maximum isometric muscle strength of the Quadriceps femoris muscle will be measured with a dynamometer (Lafayette Instrument Company, Lafayette, Indiana).
Body fat ratio | 5-10 minutes
  Body fat ratio will be evaluated by bioelectrical impedance analysis. Tanita Body Fat Analyzer (model TBF 300, Tokyo, Japan) will be used during the analysis.
Lean body weight | 5-10 minutes
  Lean body weight will be evaluated by bioelectrical impedance analysis. Tanita Body Fat Analyzer (model TBF 300, Tokyo, Japan) will be used during the analysis.
Fat weight | 5-10 minutes
  Fat weight will be evaluated by bioelectrical impedance analysis. Tanita Body Fat Analyzer (model TBF 300, Tokyo, Japan) will be used during the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldberg DJ, Avitabile CM, McBride MG, Paridon SM. Exercise capacity in the Fontan circulation. Cardiol Young. 2013 Dec;23(6):824-30. doi: 10.1017/S1047951113001649. PMID 24401254
- [Background] Chen CA, Chen SY, Chiu HH, Wang JK, Chang CI, Chiu IS, Chen YS, Lu CW, Lin MT, Lue HC, Hua YC, Wu MH. Prognostic value of submaximal exercise data for cardiac morbidity in Fontan patients. Med Sci Sports Exerc. 2014 Jan;46(1):10-5. doi: 10.1249/MSS.0b013e31829f8326. PMID 23846156
- [Background] d'Udekem Y. Cardiorespiratory Fitness, Not the Severity of the Condition, Dictates Late Outcomes After Fontan Procedures. J Am Coll Cardiol. 2017 Jun 6;69(22):2745-2747. doi: 10.1016/j.jacc.2017.03.581. No abstract available. PMID 28571640
- [Derived] Tekerlek H, Saglam M, Kucukdagli AC, Aykan HH, Vardar-Yagli N, Calik-Kutukcu E, Inal-Ince D, Karagoz T. Assessment of exercise capacity using field walking tests in patients after the Fontan procedure: A case-control study. Heart Lung. 2023 Jul-Aug;60:66-73. doi: 10.1016/j.hrtlng.2023.02.022. Epub 2023 Mar 14. PMID 36924606